CLINICAL TRIAL: NCT01271478
Title: Effect of Telmisartan and Captopril on Systemic Inflammation of Patients on Hemodialysis
Brief Title: Use of Telmisartan and Captopril in Inflammation of Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Alfonso Martín Cueto Manzano, Head, Medical Research Unit of Renal Diseases, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIS/IMSS/PROT/G09/739; Registry CLIS (Registry Identifier: R-2009-1301-83)
Record Dates: First submitted 2011-01-03; First posted 2011-01-06 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Inflammation; End-stage Renal Disease
Keywords: inflammation; telmisartan; captopril; hemodialysis
MeSH Terms: conditions — Inflammation; Kidney Failure, Chronic | interventions — Captopril; Telmisartan; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Telmisartan plus Captopril (Experimental): captopril 50 mg/day (1 tablet of 25 mg orally twice a day) plus telmisartan 80 mg/day (1 tablet of 40 mg orally twice a day)
  Interventions: Drug: Telmisartan plus Captopril
- Telmisartan plus Placebo (Experimental): telmisartan 80 mg/day (1 tablet of 40 mg orally twice a day) plus 1 tablet of placebo orally twice a day
  Interventions: Drug: telmisartan plus placebo
- Captopril plus Placebo (Experimental): patients received captopril 50 mg/day (1 tablet of 25 mg orally twice a day) plus 1 tablet of placebo orally twice a day
  Interventions: Drug: captopril plus placebo
- Placebo (Placebo Comparator): 2 tablets of placebo orally twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: captopril plus placebo — This group will receive captopril 50 mg/day (1 tablet of 25 mg orally twice a day) plus 1 tablet of placebo orally twice a day
  Other Names: Capotena
  Arms: Captopril plus Placebo
Drug: telmisartan plus placebo — Patients of this group will receive telmisartan 80 mg/day (1 tablet 40 mg orally twice a day) plus 1 tablet of placebo twice a day
  Other Names: micardis
  Arms: Telmisartan plus Placebo
Drug: Telmisartan plus Captopril — Patients of this group will receive captopril 50 mg/day (1 tablet 25 mg orally twice a day) plus telmisartan 80 mg/day (1 tablet 40 mg orally twice a day)
  Other Names: Capotena; Micardis
  Arms: Telmisartan plus Captopril
Drug: Placebo — Patients in this group will receive 2 tablets of placebo (starch) twice a day.
  Other Names: Starch
  Arms: Placebo

SUMMARY:
The aim of this study was to compare the dual use of telmisartan and captopril vs the individual use of such drugs and placebo on the systemic inflammation of patients on hemodialysis (HD).

DETAILED DESCRIPTION:
Once included, patients will be randomly allocated (by a computer-generated randomization list) to one of the following groups: group 1 will receive Captopril, group 2 Telmisartan, group 3 Captopril plus Telmisartan, and group 4 Placebo. Drugs will be provided as tablets during a period of 3 months. All patients will have 3 HD sessions per week, with the same kind of single-use dialysis membrane and dialysate Monthly visits will be scheduled for clinical and biochemical evaluations. A blood sample will be taken at baseline and every month for measurement of complete blood count, urea, creatinine, glucose, albumin, lipids, and electrolytes (measured by usual methods). In serum samples at 0, 1 and 3 months, tumor necrosis factor alpha (TNF-α) and interleukin 6 (IL-6) concentrations will be measured by ELISA using high sensitivity kits. Additionally, in the same serum samples, C-reactive protein (CRP) concentrations will be measured by nephelometry using high sensitivity kits. All laboratory measurements, including inflammation markers, will be performed in the Central Laboratory (Hospital de Especialidades, Centro Médico Nacional de Occidente), by the same personnel blinded to patient's details.

Treatment compliance will be recorded by counting tablets left in the container at the end of each monthly visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ≥2 months on hemodialysis
* Arteriovenous fistula as vascular access
* Endorsement of informed consent

Exclusion Criteria:

* Inflammatory cause of ESRD
* Liver disease, cancer, AIDS
* Any infectious disease 2 months before the study
* Failed kidney graft
* Hypersensitivity to angiotensin converting enzyme inhibitors or angiotensin receptor blockers
* Arterial hypotension
* Pregnancy
* Treatment with antibiotics, non-steroidal anti-inflammatory drugs, steroids, immunosuppressives, statins, ACE inhibitors or ARB 3 months previous to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of TNF-a, IL-6 and CRP | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso M. M Cueto-Manzano, MD, MSc, PhD, Study Chair — Unidad de Investigación Médica en Enfermedades Renales, Hospital de Especialidades, CMNO, IMSS
Locations (1):
- Hospital de Especialidades, CMNO, IMSS, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Ordaz-Medina SM, Gonzalez-Plascencia J, Martin del Campo F, Rojas-Campos E, Montanez-Fernandez JL, Espinoza-Gomez F, Cueto-Manzano AM. Is systemic inflammation of hemodialysis patients improved with the use of enalapril? Results of a randomized, double-blinded, placebo-controlled clinical trial. ASAIO J. 2010 Jan-Feb;56(1):37-41. doi: 10.1097/MAT.0b013e3181c1d830. PMID 20051840